CLINICAL TRIAL: NCT04819698
Title: Evaluation of Perioperative Cardiac Complications in Noncardiac Surgery in Tibet Autonomous Region in China：the Incidence, Risk Factors and Cardiac Troponin Monitoring
Brief Title: Perioperative Cardiac Complications in Noncardiac Surgery in Tibet, China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Tibet Autonomous Region People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LZJ003
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Perioperative Cardiac Complications
MeSH Terms: interventions — Troponin I

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Troponin I (cTnI ) monitoring — cTnI will be measured at baseline prior to surgery, as well as on 1h,12h, 24h and 72h after surgery for each patient in study B.

SUMMARY:
This observational study will describe the incidence and risk factors of perioperative cardiac complications (PCCs) in patients undergoing non-cardiac surgery in Tibet Autonomous Region. And perioperative troponin monitoring will be implemented in these population.

DETAILED DESCRIPTION:
Background: Worldwide, more than 300 million major noncardiac surgeries are performed every year and the number is increasing continuously. Perioperative cardiac complications (PCCs) are the first causes of morbidity and mortality within 30 days after noncardiac surgery which result in prolonged length of stay, increased health care costs and poorer prognosis. Several preoperative factors such as advanced age, obesity, coronary artery disease, heart failure (HF), cerebrovascular disease, diabetes mellitus, and renal dysfunction has been confirmed strongly associated with PCCs, as well as some intraoperative factors (hypotension and hypoxemia), and postoperative factors (pain and bleeding). And more than 3% patients undergoing noncardiac surgery are estimated to suffer a myocardial injury after noncardiac surgery (MINS), defined as elevated postoperative troponin measurement without the requirement of an ischemic feature. Many of the patients with MINS does not fulfill the conventional clinical diagnosis of myocardial infarction (e.g., ischemic symptom, ischemic electrocardiography finding). However, the prognosis of MINS is very poor. Therefore, cardiac troponin levels need to be monitored in high-risk patients to avoid misdiagnosis and taking the opportunity of secondary prophylactic measures and following-up.

Tibet Autonomous Region in China is located in a low-oxygen, low-pressure area, with the average altitude of more than 4000 meters. Polycythemia and hyperlipemia are common in native patients there, with increased prostaglandin, faster basal heart rate, higher blood pressure and higher myocardial oxygen consumption and restricted cardiac reserve function comparing to patients from plains areas. The mismatch between oxygen supply and demand could aggravate in the perioperative period, which is the prominent pathogenesis on PCCs. Accordingly, the risk of PCCs may rise remarkably in the high-altitude and hypoxia region. Not only that, the incidence characteristics and risk factors of PCCs in noncardiac surgery could be also partially different from those in flat area in China. However, the relevant data are currently blank.

Aim: To evaluate the incidence of PCCs, the risk indicators and the value of cardiac troponin monitoring for patients undergoing noncardiac surgery in Tibet Autonomous Region in China, allowing a better assessment and optimizing of the patients there.

Methodology: The study consists of two sub studies. Sub study A: Risk factors of PCCs in patients undergoing non-cardiac surgery in Tibet Autonomous Region. Sub study B: Implement perioperative cardiac troponin I (cTnI) monitoring.

Study A: 600 patients over 50 years old undergoing elective major noncardiac surgery in Tibet Autonomous Region People's Hospital will be included and followed for 30 days after surgery for the occurrence of PCCs and other major adverse events. Patients will receive a standardized evaluation, including preoperative historical, laboratory, and physiologic assessment. Perioperative information will also be collected, including type of surgery, anesthetic management, intraoperative transfusion, postoperative complications, etc. PCCs are defined as acute coronary syndrome (ACS), HF, new-onset severe arrhythmia, nonfatal cardiac arrest, and cardiac death.

Study B: 100 patients over 50 years old undergoing major noncardiac surgery in Tibet Autonomous Region People's Hospital will be included. Clinical data including demographics, preoperative evaluation, surgical invasiveness, ASA grade, anesthetic management, and other relevant perioperative information. The investigators will measure cTnI at baseline prior to surgery, as well as on 1h,12h, 24h and 72h after surgery for each patient. MINS will be defined if a rise of cTnI with an absolute value above the 99th percentile upper reference is detected, and then a clinical evaluation, 12-lead ECG and even coronary angiography (if needed) will be performed to adjudicate the occurrence of PCCs. The incident of MINS and the value of cTnI monitoring for early diagnosis of PCCs will be assessed for patients undergoing noncardiac surgery in Tibet Autonomous Region.

Potential Significance: This study will generate major scientific implications by contributing to closing current knowledge gaps concerning the incidence and risk factors of PCCs, as well as the value of cTnI monitoring for patients undergoing noncardiac surgery in Tibet Autonomous Region. This knowledge will have important clinical implications in the high-attitude area leading to a better optimization of the perioperative management.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 years or older；
* Undergoing intermediate to high-risk elective noncardiac surgery .

Exclusion Criteria:

* Emergency surgery;
* Local anesthesia;
* Low-risk surgery;
* ASA classification V or VI

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 50 years or older undergoing intermediate to high-risk elective noncardiac surgery.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Perioperative cardiac complications | Participants will be followed for 30 days after surgery
  Perioperative cardiac complications are defined as acute coronary syndrome (ACS), heart failure, new-onset severe arrhythmia, nonfatal cardiac arrest, and cardiac death. ACS included ST-elevation myocardial infarction (STEMI) and non-ST-elevation acute coronary syndrome (NSTE-ACS). NSTE-ACS could be further subdivided into non-ST-elevation myocardial infarction and unstable angina according to the cardiac biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zhu Q, Duan H, Liu Z, Li Y, Zhang Y, Labaciren, Shen L, Huang Y. The incidence and risk factors of perioperative cardiac complications in noncardiac major surgery in high-altitude areas: A prospective trial in Tibet autonomous region, China. Front Cardiovasc Med. 2023 Apr 3;10:1158711. doi: 10.3389/fcvm.2023.1158711. eCollection 2023. PMID 37077733